CLINICAL TRIAL: NCT05128513
Title: Delipid Extracorporeal Lipoprotein Filter From Plasma (DELP) for Acute Hemorrhagic Stroke: a Prospective, Random, Open-label, Blind-endpoint, Multi-centre Study
Brief Title: Delipid Extracorporeal Lipoprotein Filter From Plasma (DELP) for Acute Hemorrhagic Stroke
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding issues from sponsors
Sponsor: General Hospital of Shenyang Military Region (Other)
Responsible Party: Principal Investigator, Hui-Sheng Chen, Head of Neurology, General Hospital of Shenyang Military Region
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Y (2021) 38
Record Dates: First submitted 2021-10-29; First posted 2021-11-22 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Hemorrhagic Stroke
MeSH Terms: conditions — Hemorrhagic Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DELP (Experimental): Delipid Extracorporeal Lipoprotein filter from Plasma (DELP) is a non-pharmacological therapy for acute stroke, which is approved by China Food and Drug Administration
  Interventions: Device: DELP
- control group (No Intervention)

INTERVENTIONS:
Device: DELP — The blood was pumped into the PCS2 plasma separator through one side of the forearm vein. The plasma was separated by pump and then sent to the DELP system (Shanghai Jiangxia Blood Technology Co.). After purification, the plasma was returned to the patient via another forearm vein. The total treatment plasma volume was 800-1,000 mL; the anticoagulant 4% sodium citrate dehydrate solution with a ratio of 1:16 to plasma, was dropped before pumping. To prevent hypocalcemia, 500 mg CaCl2 diluted with 250 mL physiological saline was infused at a rate of 150 mL/h, in the first cycle of the returning blood transfusion.
  Arms: DELP

SUMMARY:
Delipid Extracorporeal Lipoprotein filter from Plasma (DELP) has been found to improve neurological function and life ability of AIS patients and approved for the treatment of AIS by China Food and Drug Administration (CFDA). A recent study imply that the neuroprotective effect of DELP involved multiple neuroprotective mechanism such as anti-inflammation, free radical scavenging, and decreasing MMP-9. Based on the multiple mechanisms, the investigator argues that DELP may exert neuroprotective effect on acute cerebral hemorrhage (ACH). In this context, the prospective, random, open-label, blind-endpoint, multi-centre study is designed.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-80;
* Spontaneous cerebral hemorrhage;
* Deep supratentorial intracerebral hemorrhage (basal ganglia) with hematoma volume 5-40ml, or supratentorial lobar hemorrhages with hematoma volume 5-30ml;
* NIHSS: 6-20;
* Time from onset to DELP: 6-48 hours;
* Premorbid mRS 0 or 1;
* Signed informed consent;

Exclusion Criteria:

* Secondary cerebral hemorrhage (secondary to trauma, tumor, vascular malformation, hemorrhage transformation of ischemic stroke, etc.);
* Comatose patients on admission (GCS score 3-8 on the Glasgow Coma Scale);
* Patients with intracerebral hemorrhage ruptured into the ventricle, which should be treated by surgery;
* Planed surgery;
* Severe hepatic or renal dysfunction, increase in ALT or AST (more than 2 times of upper limit of normal value), increase in serum creatinine (more than 1.5 times of upper limit of normal value) or requiring dialysis;
* Severe hypertension (systolic blood pressure over 200mmHg or diastolic blood pressure over 110 mmHg), or hypotension (systolic blood pressure below 90mmHg or diastolic blood pressure below 60 mmHg);
* Previous allergy to heparin or calcium;
* Life expectancy is less than 6 months due to comorbidity
* Infected at the venipuncture site
* hypoproteinemia;
* Unsuitable for this clinical studies assessed by researcher.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 356 (Estimated)
Dates: Start 2022-01-14 (Actual); Primary Completion 2026-02-08 (Estimated); Study Completion 2026-02-08 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with modified Rankin Score 0 to 2 | Day 90
  the minimum and maximum values of modified Rankin Score are 0 and 6, respectively; higher score mean a worse outcome

SECONDARY OUTCOMES:
Proportion of patients with modified Rankin Score 0 to 1 | Day 90
  the minimum and maximum values of modified Rankin Score are 0 and 6, respectively; higher score mean a worse outcome
distribution of modified Rankin Score | Day 90
  the minimum and maximum values of modified Rankin Score are 0 and 6, respectively; higher score mean a worse outcome
Changes in National Institute of Health stroke scale (NIHSS) | 24 hours and 2 weeks
  the minimum and maximum values of NIHSS are 0 and 42, respectively; higher NIHSS mean a worse outcome
the occurence of stroke or other vascular events | Day 90
the changes in cerebral hematoma volume | 24 hours
  the hematoma volume was formulated by brain CT
the severe adverse events | 24 hours
the occurence of death due to any cause | 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurology, General Hospital of Northern Theater Command, Shenyang, China

IPD SHARING:
Plan to Share IPD: Undecided